CLINICAL TRIAL: NCT03777358
Title: A Prospective Study Comparing Three-dimensional Ultrasonography Versus Hysteroscopy in Evaluation of Uterine Cavity in Infertile Women
Brief Title: Three-dimensional Ultrasonography Versus Hysteroscopy in Evaluation of Uterine Cavity in Infertile Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hatem AbuHashim (Other)
Responsible Party: Sponsor-Investigator, Hatem AbuHashim, Professor, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: MD.18.10.99
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Three-dimensional transvaginal ultrasonography (3D-TVS): The 3D-TVS will be done by an experienced gynecological sonographer. The uterine cavity will be assessed by obtaining a mid-coronal view. Then, hysteroscopy will be performed.
  Interventions: Device: 3D-TVS

INTERVENTIONS:
Device: 3D-TVS — The 3D-TVS will be done by an experienced gynecological sonographer. The uterine cavity will be assessed by obtaining a mid-coronal view. Then hysteroscopy will be performed

SUMMARY:
Hysteroscopy has now become a gold-standard technique carried out for uterine cavity assessment in infertile women. Apart from direct visualizing of the endometrium by the naked eye, pathologies missed by other modalities of investigation can be picked up and managed appropriately. Unfortunately, the procedure itself is not free from complications e.g. perforation, cervical laceration, bleeding, limited access in cases of cervical stenosis and considered as an invasive procedure.

Two-dimensional transvaginal ultrasonography (2D-TVS)and Three-dimensional TVS (3D-TVS) are non-invasive methods for evaluating the uterine cavity. The3D-TVS is superior to 2D-TVS in identifying uterine cavity abnormalities due to its ability to obtain a view of three different planes of the uterus, which could be used to locate the position of intracavitary pathology. Reports vary regarding the diagnostic accuracy of 3D-TVS that was reported to have 41.3-81.5% sensitivity and 94.6-98.7% specificity. So it became clear that 3D-TVS is a non-invasive and safe diagnostic tool for evaluation of the uterine cavity abnormalities but its sensitivity, specificity and accuracy still a matter of debate and warrants more evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women (primary or secondary)
* Age between 18 and 40 years.

Exclusion Criteria:

* age<18 years and˃ 40 years.
* pelvic inflammatory disease.
* .Active uterine bleeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women (primary or secondary) aged between 18 and 40 years.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of 3D-TVS | At 1 week postmenstrual
  The diagnostic accuracy of 3D-TVS in comparison with hysteroscopy for evaluation of uterine cavity abnormalities in infertile women.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. FRCOG. PhD, Study Chair — Faculty of Medicine, Mansoura University; Mohamed Fekry, MSc, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Ahmadi F, Rashidy Z, Haghighi H, Akhoond M, Niknejadi M, Hemat M, Shamsipour M. Uterine cavity assessment in infertile women: Sensitivity and specificity of three-dimensional Hysterosonography versus Hysteroscopy. Iran J Reprod Med. 2013 Dec;11(12):977-82. PMID 24639723